CLINICAL TRIAL: NCT02255227
Title: Phase IIb Multicenter Randomized Comparative Study of Anti-pneumococcal Vaccine Strategy in Patients Treated With Immunosuppressants or Biotherapies for Chronic Inflammatory Bowel Disease
Brief Title: Anti-pneumococcal Vaccine Strategy in Patients Treated With Immunosuppressants or Biotherapies for CIBD
Acronym: PneumoMICI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low inclusion rates
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1308162; 2013-004609-19 (EudraCT Number)
Record Dates: First submitted 2014-09-26; First posted 2014-10-02 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Infections, Pneumococcal; Bowel Diseases, Inflammatory
Keywords: vaccination; randomized; anti-pneumococcal; Pneumo 23; Prevenar 13; Chronic Inflammatory Bowel Disease
MeSH Terms: conditions — Pneumococcal Infections; Inflammatory Bowel Diseases | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 dose Prevenar13 and 1 dose PSV23 (Active Comparator): one dose of the polysaccharide vaccine, Prevenar 13 at M0 and one dose of polysaccharide vaccine, Pneumo 23 at M4
  Interventions: Biological: Prevenar 13; Biological: Pneumo 23
- 2 doses Prevenar13 and 1 dose PSV23 (Experimental): one dose of the polysaccharide vaccine, Prevenar 13 at M0, one dose of the polysaccharide vaccine, Prevenar 13, at M2 and one dose of polysaccharide vaccine, Pneumo 23 at M4
  Interventions: Biological: Prevenar 13; Biological: Pneumo 23

INTERVENTIONS:
Biological: Prevenar 13 — one dose for arm 1 and 2 doses for arm 2
Biological: Pneumo 23 — one dose

SUMMARY:
This is a multicenter, prospective, randomized, open study comparing two anti-pneumococcal vaccination strategies in patients with Chronic Inflammatory Bowel Disease (CIBD) treated by immunosuppressants and/or biotherapies. At present such patients are poorly protected by anti-pneumococcal vaccination. In addition, vaccination efficacy in this type of patient is much weaker than in the general population. There are two types of anti-pneumococcal vaccines: firstly a polysaccharide, Pneumo23® (PSV-23®) vaccine and secondly a conjugate, Prevenar13® vaccine. New recommendations have just been issued by the HSCP advising immunocompromised patients to follow a vaccination plan combining one dose of Prevenar13® followed by one dose of PSV-23® after an interval of two months. In the case of young children infected with HIV, the recommendation is to multiply doses of Prevenar13® before the PSV-23® injection to improve vaccine efficacy in these immunocompromised patients.

Our study aims to identify an optimal vaccination strategy for immunocompromised CIBD patients by combining use of a conjugate vaccine, Prevenar13® and a polysaccharide vaccine, PSV-23®. We will compare the use of one or two doses (M0 +/- M2) of Prevenar13® combined with a later PSV-23® injection (M4) on vaccination immunogenicity measured by antibody titer against at least nine of the thirteen pneumococcal serotypes contained in Prevenar13®. We also want to evaluate the immunological impact of these different strategies in their capacity to stimulate a memory B anti-pneumococcal response more effectively. With this aim, we are studying all immunological functional aspects of the antibodies and B lymphocytes induced by the two vaccine strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have given their written consent in a free and informed consent
* Patient followed for inflammatory bowel disease (Crohn's disease, ulcerative colitis or indeterminate colitis), and treated for at least 3 months by immunosuppressive therapy and /or biotherapies and in clinical remission for at least 3 months
* Patient agreeing to participate in the study throughout its duration and accepting the procedures related to the study
* Contraception that the investigator judges effective for the first 12 months of the trial, with a negative pregnancy test
* Women not planning to become pregnant in the 12 months following inclusion (M0)
* Patient with social coverage

Exclusion Criteria:

* Patients vaccinated against pneumo23 for less than 5 years
* Other vaccination during the month before inclusion
* Patient develops a febrile illness (at least 37 ° C 5 measured orally) or acute infection in the week before vaccination
* The patient has a flare up of IBD the day of vaccination (Harvey-Brasdshaw score of at least 6 or CDAI > 220 for Crohn's disease or Mayo Clinic score of at least 4 for UC and indeterminate colitis)
* Patients with an ongoing pregnancy the day of vaccination
* Patient with a known history of neuropathy as Guillain-Barré syndrome.
* Patients with known infection with HIV and / or HBV (HBsAg positive) and / or HCV
* Patient with other severe immune deficiency
* Patients who received immunoglobulin infusions of blood products, or of monoclonal antibodies (except anti-TNF) in the 3 months prior to vaccination
* Patient institutionalized, or deprived of liberty administrative or judicial
* Patients treated without immunosuppressive therapy or biotherapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-04-13 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
number of patients with anti-pneumococcal immunogenicity | month 5
  Measured the serologies against serotypes to Prevenar 13. Serotype to be measured are 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A 19 F and 23F using the ELISA method

SECONDARY OUTCOMES:
Number of patients with local and/or general reaction | Months 1, 3 and 5
  self monitoring diary
Number of patients with inflammatory disease activity | Months 1, 3, 4, 5, 12, 18, 36
  by clinic score HBI or CDAI or Mayo
Factors implicated in anti-pneumococcal vaccination efficacy | Month 0
  questionnaire
number of patients with serotype coverage of PSV-23 | Months 5, 12, 18 and 36
  Measured the serologies against serotypes to Pneumo 23. Serotype to be measured are serotypes 10 and 15 using the ELISA method

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Roblin, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (8):
- France (8):
  - CHU Amiens-Picardie, Amiens
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Saint-Eloi, Montpellier
  - Hôpital de l'Archet II, Nice
  - APHP - Hôpital Cochin, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Charles Nicolle, Rouen
  - CHU de Saint-Etienne, Saint-Etienne